CLINICAL TRIAL: NCT02936726
Title: The Healthy Staff Initiative Study: Examining Exercise, Health Coaching and Meditation for University Employees: a Randomized Trial
Brief Title: Examining Exercise, Health Coaching and Meditation for University Employees
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment Completed
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Shalini Moonsammy Persaud, PhD. Canditate, York University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU 2016 - 121
Record Dates: First submitted 2016-10-12; First posted 2016-10-18 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Motor Activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise and Health Coaching (Active Comparator): Walking exercise protocol program, carried out by themselves, over 12 weeks.
  Health Coach addresses various topics with participant, half-hour sessions on a weekly (12 sessions)
  Interventions: Behavioral: Exercise and Health Coaching
- Exercise, Health Coaching and Meditation (Experimental): Walking exercise protocol program, carried out by themselves, over 12 weeks.
  Health Coach addresses various topics with participant, half-hour sessions on a weekly (12 sessions)
  Mindfulness Meditation intervention will incorporate varied types of MBI techniques 3 times per week for 12 weeks, during work hours and/or during their time on campus (after work hours).
  Interventions: Behavioral: Exercise, Health Coaching and Meditation

INTERVENTIONS:
Behavioral: Exercise, Health Coaching and Meditation — Comparing Exercise, Health Coaching and Meditation In Combination
  Arms: Exercise, Health Coaching and Meditation
Behavioral: Exercise and Health Coaching — Comparing Exercise and Health Coaching Alone
  Arms: Exercise and Health Coaching

SUMMARY:
There is evidently great potential in implementing workplace health promotion programs, but more randomized trials are needed to determine which interventions are worksite-effective in helping to decrease inactive behaviors and increase engagement in healthy lifestyle activities. For employers, it could mean improving the health and productivity of employees. For workers, especially those in physically and/or psychologically demanding positions, it could mean developing strength, muscular endurance and agility to reduce musculoskeletal pain while developing the stress reduction skills that reduce long-term sickness and absenteeism risks. While changing behavior in a complex workplace is, as seen in multiple studies, difficult due to the need to change workplace and organizational culture between employers and employees, this study aims to identify the effectiveness of workplace interventions in relation to counseling for university employees to increase overall work fitness without affecting any hierarchal interactions at the work site. Simply put, the investigators will examine the benefits of a workplace exercise and mindfulness (two-prong) intervention (in combination) vs. a group who just receive a workplace exercise intervention. Both interventions will be guided by health coaches. Given the limited research with health coaching and workplace interventions for university workers, the aim is to contribute to a developing research literature. This study is geared to engage university employees at their workplace over a 3 month period. Participants will be assessed through pre and post physical and psychological measures and will also undergo semi-structured interviews (SSI).

DETAILED DESCRIPTION:
There is evidently great potential in implementing workplace health promotion programs, but more randomized trials are needed to determine which interventions are worksite-effective in helping to decrease inactive behaviors and increase engagement in healthy lifestyle activities. For employers, it could mean improving the health and productivity of employees. For workers, especially those in physically and/or psychologically demanding positions, it could mean developing strength, muscular endurance and agility to reduce musculoskeletal pain while developing the stress reduction skills that reduce long-term sickness and absenteeism risks. While changing behavior in a complex workplace is, as seen in multiple studies, difficult due to the need to change workplace and organizational culture between employers and employees, this study aims to identify the effectiveness of workplace interventions in relation to counseling for university employees to increase overall work fitness without affecting any hierarchal interactions at the work site. Simply put, the investigators will examine the benefits of a workplace exercise and mindfulness (two-prong) intervention (in combination) vs. a group who just receive a workplace exercise intervention. Both interventions will be guided by health coaches. Given the limited research with health coaching and workplace interventions for university workers, the aim is to contribute to a developing research literature. This study is geared to engage university employees at their workplace over a 3 month period. Participants will be assessed through pre and post physical and psychological measures and will also undergo semi-structured interviews (SSI). The investigators hypothesize that making available these various fitness and well-being programs for university employees will effectively improve their overall fitness (peak VO2) and psychological health (stress, depression, anxiety, work satisfaction), making them more efficient, positive and work-productive. Specifically, the investigators hypothesize that the exercise and mindfulness meditation group will demonstrate significant improvements when compared to the group solely receiving exercise-oriented health coaching. Improvements will be seen across all measures of physical (such as VO2 peak and BMI) and psychological (such as depression, stress, anxiety, work-life balance) function and will be sustained at 3 month follow-up, indicating a more effective means of initiating fitness at the workplace

ELIGIBILITY:
Inclusion Criteria:

* Employees at York University;
* fluency in English;
* provision of informed consent

Exclusion Criteria:

* currently engaged in regular exercise programs or routines which meet or exceed the Canadian Physical Activity Guidelines
* neurological or musculoskeletal co-morbidities inhibiting participation in exercise program
* > 65 years old;
* medical history of cardiovascular diseases such as CAD and CHF, uncontrolled hypertension
* currently engaged in a mindfulness meditation program or meditative practice at advanced levels;
* not in possession of a smartphone (android/i-phone)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
VO2 Peak | Baseline, 12 weeks and 24 weeks
  Assess changes in VO2 peak over time

SECONDARY OUTCOMES:
Psychological Questionnaires | Baseline, 12 weeks and 24 weeks
  Assess changes over time

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Moonsammy Persaud, PhD (cand), Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data is analyzed as group data

REFERENCES:
- [Background] Jakobsen MD, Sundstrup E, Brandt M, Kristensen AZ, Jay K, Stelter R, Lavendt E, Aagaard P, Andersen LL. Effect of workplace- versus home-based physical exercise on pain in healthcare workers: study protocol for a single blinded cluster randomized controlled trial. BMC Musculoskelet Disord. 2014 Apr 7;15:119. doi: 10.1186/1471-2474-15-119. PMID 24708570
- [Background] van Berkel J, Boot CR, Proper KI, Bongers PM, van der Beek AJ. Effectiveness of a worksite mindfulness-based multi-component intervention on lifestyle behaviors. Int J Behav Nutr Phys Act. 2014 Jan 27;11:9. doi: 10.1186/1479-5868-11-9. PMID 24467802
- [Background] Marshall AL. Challenges and opportunities for promoting physical activity in the workplace. J Sci Med Sport. 2004 Apr;7(1 Suppl):60-6. doi: 10.1016/s1440-2440(04)80279-2. PMID 15214603